CLINICAL TRIAL: NCT01382836
Title: The Role of Epigenetics in Inner City Asthma (ICAC-15)
Brief Title: The Role of Epigenetics in Inner City Asthma
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT ICAC-15
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA, RNA, serum, and plasma specimens
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Black inner city children with persistent asthma
- Black inner city non-atopic healthy children

SUMMARY:
As part of ongoing efforts to determine the causes of asthma and the progression of the disease, this study will gather data to explore the interaction of genetic and environmental factors in the cause and severity of asthma in inner city children.

DETAILED DESCRIPTION:
Asthma is a complex, heritable disease that affects more than 11.2% of the U.S. population, which represents approximately 9 million children and 23 million adults. It is thought that asthma may be caused by the interaction of multiple genetic factors, such as whether a parent or sibling has asthma, and environmental factors, such as living in an inner city. Studying DNA from people who have asthma and those who do not have asthma may help us better understand the importance of those genes and how they are involved in asthma severity and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

-Black inner city children with or without asthma.

Control Subjects:

-Black males and females ages 6 to 12 years, inclusive, at Recruitment;

* Who do not have a diagnosis of asthma by a physician;
* Who do not have a diagnosis of atopic dermatitis by a physician;
* Who have an FEV1 ≥ 85% predicted;
* With no positive prick skin-tests to any of a panel of indoor and outdoor allergens;
* With no current asthma as determined by the Respiratory Health Questionnaire (RHQ);
* With no current chronic rhinitis/sinusitis as determined by the RHQ;
* Whose primary place of residence is in one of the pre-selected recruitment census tracts that contains at least 15% of households below the U.S. government poverty level;
* Who are able to perform spirometry (according to the Epigenetics Manual of Operations criteria);
* Whose parent or legal guardian is willing to sign the written Informed Consent prior to initiation of any study procedure;
* Who are willing to sign the assent form, if age appropriate.

Asthmatic Participants:

* Black males and females ages 6 to 12 years, inclusive, at Recruitment;
* Who have a diagnosis of asthma by a physician;
* Who are currently receiving long-term asthma control therapy and either have symptoms consistent with persistent asthma (criterion 3a) or have evidence of uncontrolled disease (criterion 3b); or who are not currently receiving long-term asthma control therapy and have symptoms consistent with persistent asthma (criterion 3a) and have evidence of uncontrolled disease (criterion 3b);
* Evidence of persistent asthma as defined by the National Asthma Education and Prevention Program (NAEPP) Expert Panel Report 3: Guidelines for the Diagnosis and Management of Asthma (NHLBI 2007), which includes at least one of the following criteria:

  * Asthma symptoms 3 or more days per week during the last two weeks;
  * Sleep disturbed due to asthma at least 3 times in the past month;
  * Albuterol use (Metered Dose Inhaler or nebulizer) for quick relief at least 8 times in the past two weeks, not including use as a preventive for exercise.
* Evidence of uncontrolled disease as defined by at least one of the following criteria:

  * Two or more asthma-related unscheduled visits to an emergency department (ED), urgent care (UC), or clinic in the previous 6 months;
  * One or more asthma-related overnight hospitalizations in the previous 6 months.
* With physiologic evidence of reversible airflow obstruction or airway hyperresponsiveness:

  * FEV1 < 85% predicted or FEV1/FVC ratio < 0.85 with a bronchodilator response ≥ 10% FEV1;
  * Positive methacholine challenge (PC20 < 8 mg/ml) for those individuals who have either:
  * Normal airflow (FEV1 ≥ 85% predicted and FEV1/FVC ratio ≥ 0.85);
  * Airflow obstruction with a bronchodilator response < 10% FEV1.
* With a positive prick skin-test to at least one of the panel of indoor aeroallergens (i.e. dust mite, cockroach, mold, cat, dog, rat, mouse);
* Whose primary place of residence is in one of the pre-selected recruitment census tracts that contains at least 15% of households below the U.S. government poverty level;
* Who are able to perform spirometry;
* Whose parent or legal guardian is willing to sign the written Informed Consent prior to initiation of any study procedure;
* Who are willing to sign the assent form, if age appropriate.

Exclusion Criteria:

* Who have a sibling already enrolled in the study (i.e. one individual from each family is permitted to participate [case or control], though samples will be collected from parents and siblings);
* Who have received systemic prednisone (or equivalent) during the 30 days prior to the screening visit;
* Who have received systemic prednisone (or equivalent) for > 15 days out of the past 60 days prior to the screening visit;
* Who are pregnant or lactating;
* With acute sinusitis, chest infection, or ear infection that required treatment with antibiotics within 30 days of the screening visit;
* Who are currently participating in another asthma-related pharmaceutical study or intervention study or who have participated in another asthma-related pharmaceutical study or intervention study in the month prior to the screening visit;
* Who are currently receiving or have received hyposensitization therapy to any allergen in the past year prior to the screening visit;
* Who have the presence of the following chronic medical conditions: cardiac condition requiring daily medication, seizure disorder requiring daily medication, obvious severe mental retardation that prohibits the subject from answering questions or following instructions, cystic fibrosis, immune deficiency, diabetes, allergic bronchopulmonary aspergillosis, or any other chronic medical condition at the discretion of the study physician. (Exceptions: Attention deficit disorder with or without hyperactivity; iron deficiency anemia; gastroesophageal reflux disease; otitis media (ear infections); sinusitis; allergic rhinitis);
* Who do not speak and understand English;
* Whose caretaker does not speak and understand English.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Black inner city children with:1.)persistent asthma and 2.) without asthma.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Global DNA methylation patterns in PBMCs isolated from the persistent asthmatics and non-atopic healthy controls | 24 months

SECONDARY OUTCOMES:
Global DNA methylation patterns in nasal epithelial cells | 24 months
DNA methylation patterns in PBMCs isolated from the parent(s) and/or siblings | 24 months
Gene expression profiles of RNA extracted from PBMCs and nasal epithelial cells of the persistent asthmatics and non-atopic healthy controls | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: David Schwartz, MD, Study Chair — National Jewish Health; Andrew Liu, MD, Study Chair — National Jewish Health
Locations (6):
- United States (6):
  - National Jewish Health, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Boston University School of Medicine, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Result] Yang IV, Pedersen BS, Liu A, O'Connor GT, Teach SJ, Kattan M, Misiak RT, Gruchalla R, Steinbach SF, Szefler SJ, Gill MA, Calatroni A, David G, Hennessy CE, Davidson EJ, Zhang W, Gergen P, Togias A, Busse WW, Schwartz DA. DNA methylation and childhood asthma in the inner city. J Allergy Clin Immunol. 2015 Jul;136(1):69-80. doi: 10.1016/j.jaci.2015.01.025. Epub 2015 Mar 11. PMID 25769910
- See also: NIAID Programs on Asthma in the Inner City — http://www.niaid.nih.gov/topics/asthma/research/Pages/innerCity.aspx#icac